CLINICAL TRIAL: NCT05377255
Title: A Phase 1, Open Label, Randomized Study to Investigate the Pharmacokinetics and Safety of Multiple Doses of Intranasal Naloxone in Healthy Adult Participants
Brief Title: Pharmacokinetics (PK) and Safety of Multiple Doses of Intranasal Naloxone in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EBS-NAR-001
Record Dates: First submitted 2022-03-11; First posted 2022-05-17 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Opioid Overdose
Keywords: NARCAN; Opioid Overdose; Naloxone; Intranasal
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Interventional Therapy (Other): Subjects will first receive 4 doses of 4 mg each (total: 16 mg) of naloxone through the AP003 device (Arm 1) before the washout period.
  Interventions: Combination Product: 16 mg naloxone AP003; Combination Product: 8 mg naloxone NARCAN Nasal Spray
- Arm 2 Reference Therapy (Other): Subjects will first receive 2 doses of 4 mg each (total: 8 mg) of the naloxone through the NARCAN Nasal Spray device (reference therapy, Arm 2) before the washout period.
  Interventions: Combination Product: 16 mg naloxone AP003; Combination Product: 8 mg naloxone NARCAN Nasal Spray

INTERVENTIONS:
Combination Product: 16 mg naloxone AP003 — 4 doses of 4 mg each (total: 16 mg) of naloxone through the AP003 device
Combination Product: 8 mg naloxone NARCAN Nasal Spray — 2 doses of 4 mg each (total: 8 mg) of the naloxone through the NARCAN Nasal Spray device

SUMMARY:
This study will be a Phase 1, single-center, open-label, randomized cross-over study to evaluate the PK of a new AP003 device which delivers two sprays of 4 mg naloxone hydrochloride intranasally.

DETAILED DESCRIPTION:
Based on the intended AP003 product presentation there will be two devices in each carton allowing for administration of a total of 16 mg. This study is designed for subjects to receive naloxone therapy either through the AP003 device or through the currently approved NARCAN® nasal spray (4 mg) device (per label), reference therapy. After administration of the therapy patients will be followed by a 48-hour washout period before treatment crossover. Key study parameters include safety and PK. Safety evaluations will include but not limited to complete and system directed physical examinations (including signs of nasal irritation such as erythema, edema, and erosion), administration of a Brief Smell Identification Test (B-SIT), assessments of vital signs, 12 lead electrocardiogram (ECG), continuous cardiac telemetry monitoring (CCT) , clinical laboratory tests (e.g., hematology, chemistry, urinalysis, pregnancy test), and evaluation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Are able to consent and freely provide informed consent.
* Females and males 18-55 years of age, inclusive.
* Have a body mass index (BMI) less than or equal to 34.0 kg/m2.
* Generally healthy, in the opinion of the Investigator, based on medical history, physical examination, vital signs, screening laboratory assessments and 12-lead ECG evaluation.
* If female:

  1. Have a negative pregnancy test at Screening (serum pregnancy test) and before dosing at Day -1 (urine pregnancy test)
  2. Female subjects of non-childbearing potential must be:

     * Post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented FSH levels ≥40 mIU/mL; or
     * Surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy, or tubal ligation) at least 3 months prior to dosing.
  3. Women of childbearing potential who are not planning to be pregnant during the study period and who are using one of the following effective methods of contraception during the study period and for at least 30 days after last study visit:

     * Simultaneous use of hormonal contraceptive (e.g. oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device for at least 4 weeks prior to dosing (must agree to use the same contraceptive throughout the study) and condom for the male partner.
     * Simultaneous use of diaphragm or cervical cap with spermicide and condom for the male partner, started at least 21 days prior to dosing.

Exclusion Criteria:

* Subjects planning to become pregnant during the study or currently breastfeeding.
* Any acute condition, in the opinion of the Investigator, that is not fully resolved at least 4 weeks prior to baseline.
* Subject has a deviated septum, previous rhinoplasty, abnormal nasal anatomy, other nasal symptoms (i.e., blocked and/or runny nose), or other nasal surgeries (i.e., polyp removal) within 1 year, or needs to use another nasal spray product during study.
* Subject with current upper respiratory infection (URI) or has had URI within 7 days prior to screening.
* Subject has had an episode of epistaxis within 30 days prior screening or has experienced recurrent episodes of epistaxis within 1 year prior to screening.
* Subject has used any prescription or nonprescription drugs/supplements with increased risk of bleeding within 28 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug with exception of oral contraceptives. All other prescription medications, over-the-counter, and natural health products within 14 days or 5 half-lives prior to the first dosing.
* Subject is currently participating in another clinical study of an investigational drug or has been dosed with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Mean naloxone plasma concentration AP003 dosing periods. | PK samples taken at various timepoints over the course of Pre-dose and post-dose for 12 hours.
  The mean naloxone plasma concentration during the two AP003 dosing periods.
Mean naloxone plasma concentration Narcan dosing periods | PK samples taken at various timepoints over the course of Pre-dose and post-dose for 12 hours.
  The mean naloxone plasma concentration during the two Narcan dosing periods.
Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAE) | Through end of study visit (within 7 days after second dose)
  Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAE) by treatment thru End of Study Visit (within 7 days after 2nd dose).
Incidence of abnormal vital signs | Through end of study visit (within 7 days after second dose)
  Incidence of abnormal vital signs (heart rate, blood pressure, and respiration rate) by treatment thru End of Study Visit (within 7 days after 2nd dose).
Incidence of clinically significant ECG | Through end of study visit (within 7 days after second dose)
  Incidence of clinically significant ECG by treatment thru End of Study Visit (within 7 days after 2nd dose).
Incidence of clinical laboratory changes | Through end of study visit (within 7 days after second dose)
  Incidence of clinical laboratory changes by treatment thru End of Study Visit (within 7 days after 2nd dose).
Incidence of adverse events of special interest (AESI) indicating of nasal irritation | Through end of study visit (within 7 days after second dose)
  Incidence of adverse events of special interest (AESI) indicating of nasal irritation (erythema, edema, and erosion) by treatment thru End of Study Visit (within 7 days after 2nd dose).
Incidence of changes in B-SIT assessment | Through end of study visit (within 7 days after second dose)
  Incidence of changes in B-SIT assessment within an AP003 period thru End of Study Visit (within 7 days after 2nd dose).

CONTACTS AND LOCATIONS:
Overall Officials: Nino Joy, MD, Study Director — Emergent BioSolutions
Locations (1):
- Syneos Health Clinical Research Services, Miami, Florida, United States